CLINICAL TRIAL: NCT03776305
Title: Pharmacokinetics of Imipenem in Critically Ill Patients With Life-threatening Severe Infections During Support With Extracorporeal Membrane Oxygenation
Brief Title: Imipenem in Critically Ill Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sutep Jaruratanasirikul, Principle Investigator, Prince of Songkla University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMIECMO2018
Record Dates: First submitted 2018-12-11; First posted 2018-12-14 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-12

CONDITIONS: Critically Ill Patients With ECMO
Keywords: pharmacokinetic; imipenem; extracorporeal membrane oxygenation
MeSH Terms: interventions — Imipenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imipenem ECMO (Experimental): 1-h infusion of 0.5 g of imipenem, q6h
  Interventions: Drug: Imipenem

INTERVENTIONS:
Drug: Imipenem — 1-h infusion of 0.5 g of imipenem diluted in 100 mL of normal saline solution, delivered via infusion pump at a constant flow rate, every 6 h. The imipenem PK studies were carried out during administration of the fourth dose of each regimen (18-24 h after the start of the regimen). Blood samples were obtained by direct venipuncture at the following times: before (time zero) and 0.25, 0.5, 0.75, 1, 2, 3, 4, 5 and 6 h after the fourth dose of each regimen.

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) has become increasingly used for lifesaving respiratory and/or cardiac failure support in critically ill patients, including those with life-threatening severe infections. This cardiopulmonary bypass device has been shown to enhance the profound pathophysiological changes in this patient population, resulting in an alteration of the pharmacokinetics (PK) of antimicrobial agents. The aim of this study was to determine the effect of ECMO on the PK of imipenem in critically ill patients supported by this cardiopulmonary bypass device.

Methods The study was conducted in critically ill patients with respiratory and/or cardiac failure and suspected severe nosocomial infections who were supported by ECMO. All patients received a 1-h infusion of 0.5 g of imipenem every 6 h and imipenem PK studies were carried out on the fourth dose of drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18 year
* Patients who diagnosed as severe sepsis
* Admitted into the ICU
* Supported with ECMO

Exclusion Criteria:

* Patients who pregnant
* Patients who have documented hypersensitivity to carbapenem

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of imipenem in plasma | 6 hour after the imipenem dose
  Individual concentration of imipenem in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Clinical Pharmacology, Department of Medicine, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Derived] Jaruratanasirikul S, Vattanavanit V, Wongpoowarak W, Nawakitrangsan M, Samaeng M. Pharmacokinetics and Monte Carlo Dosing Simulations of Imipenem in Critically Ill Patients with Life-Threatening Severe Infections During Support with Extracorporeal Membrane Oxygenation. Eur J Drug Metab Pharmacokinet. 2020 Dec;45(6):735-747. doi: 10.1007/s13318-020-00643-3. PMID 32886347